CLINICAL TRIAL: NCT02623452
Title: Pharmacokinetics, Glucodynamics, Safety, and Tolerability of a Novel Insulin Lispro Formulation in Patients With Type 1 Diabetes Mellitus on Multiple Daily Insulin Injection Therapy
Brief Title: A Study of a New Type of Insulin in Participants With Type 1 Diabetes on Insulin Injection Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in clinical strategy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15627; F3Z-FW-ITCB (Other: Eli Lilly and Company); 2015-003351-21 (EudraCT Number)
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A:Insulin Lispro Test (Experimental): Individualized doses of Insulin Lispro test formulation administered by injection under the skin once in each of 3 periods
  Interventions: Drug: Insulin Lispro
- Part A:Insulin Lispro Reference (Active Comparator): Individualized doses of Insulin Lispro reference formulation administered by injection under the skin once in each of 3 periods
  Interventions: Drug: Insulin Lispro
- Part B:Insulin Lispro Test (Experimental): Individualized doses of Insulin Lispro test formulation administered by injection under the skin with each meal for 14 days
  Interventions: Drug: Insulin Lispro
- Part B:Insulin Lispro Reference (Active Comparator): Individualized doses of Insulin Lispro reference formulation administered by injection under the skin with each meal for 14 days
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Lispro — Administered subcutaneously (SC)

SUMMARY:
The study will be conducted in participants with type1 diabetes on insulin injection therapy to investigate how the body processes a test formulation of insulin lispro and the effect of the test formulation on blood sugar levels. Side effects and tolerability will be documented. The study will be conducted in two parts (Part A and Part B) to achieve its objectives. Participants are expected to enroll in both parts.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants with type 1 diabetes mellitus (T1DM) on a stable multiple daily injection regimen with a short-acting as well as a long-acting insulin
* Have a body mass index (BMI) ranging from 18.5 to 33.0 kilogram per square meter (kg/m²), inclusive, at screening
* Have blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results acceptable for the study
* Have had no episodes of severe hypoglycemia in the past 6 months (requiring assistance in treatment by a second party)
* Have venous access sufficient to allow for blood sampling
* Have provided written consent and are willing to follow study procedures and commit to the study duration

Exclusion Criteria:

* Are currently enrolled, or have participated within the last 30 days, in a clinical trial or any other type of medical research judged to be incompatible with this study
* Have previously completed or withdrawn from this study
* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate in the study
* Had blood loss of more than 500 milliliters (mL) within the last month
* Are treated with a continuous subcutaneous insulin infusion (insulin pump)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
(Part A) Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) of Insulin Lispro | Time 0 to 5 hours post dose for each treatment on Day 1
  (Part A) PK: AUC of Insulin Lispro
(Part B) PK: AUC of Insulin Lispro | Time 0 to 5 hours post dose on Day 1 and Day 14 of study treatment
  (Part B) PK: AUC of Insulin Lispro

SECONDARY OUTCOMES:
(Part A) Pharmacodynamics (PD): AUC of Glucose Following a Meal | Time 0 to 5 hours post meal for each treatment on Day 1
  (Part A) PD: AUC of Glucose Following a Meal
(Part B) PD: AUC of Glucose Following a Meal | Time 0 to 5 hours post meal on Day1 and Day14 of study treatment
  (Part B) PD: AUC of Glucose Following a Meal

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company